CLINICAL TRIAL: NCT01744717
Title: "Estudio multicéntrico de Validez y Fiabilidad de la Escala de Conductas Indicadoras de Dolor ESCID Para Medir el Dolor en Pacientes críticos, no Comunicativos y Sometidos a ventilación mecánica"
Brief Title: Validation of "Escala de Conductas Indicadoras de Dolor" ESCID Scale for Measuring Pain in Critically Ill Patients
Acronym: ESCID-MQ
Status: Completed | Type: Observational
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital Universitario Getafe (Other); Hospital Universitario 12 de Octubre (Other); Hospital Universitario Ramon y Cajal (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital San Carlos, Madrid (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Quirón Madrid University Hospital (Other); Hospital de Cruces (Other); Hospital de Basurto (Other); Hospital Galdakao-Usansolo (Other Government); Hospital Universitario Fundación Alcorcón (Other); Hospital Universitario de Fuenlabrada (Other)
Responsible Party: Principal Investigator, Ignacio Latorre Marco, Nurse Degree, Intensive Care Unit nurse staff, Puerta de Hierro University Hospital
Other Study IDs: ESCID-02
Record Dates: First submitted 2012-11-14; First posted 2012-12-07 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Pain
Keywords: Pain; mechanical ventilation; uncommunicative; Adult ICU patients pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critically ill uncommunicative patients: Critically ill non-communicative patients, on mechanical ventilation
  Interventions: Other: Pain measurement

INTERVENTIONS:
Other: Pain measurement — Pain intensity will be measured using 2 scales based on behaviour items, the Behavioural Pain Scale (BPS) and the ESCID scale (Escala de Conductas Indicadoras de Dolor), by two independent observers , when applying two procedures registered as painful (PD) and common in clinical practice, and a non-painful procedure (PND). The measurement will be performed once per each patient and procedure.
  The procedures to be studied are the following:
  * TURNING / POSITIONING (moving side to side or up or down in bed)
  * ENDOTRACHEAL SUCTIONING (insertion of suction catheter into the endotracheal tube or tracheostomy in order to aspirate secretions)
  * NON PAINFUL PROCEDURE (Soft friction with gauze cloth on a healthy skin tissue portion, in the outer arm, forearm or anterior tibial area)

SUMMARY:
Pain is an unpleasant and important stress factor, and a potentially harmful experience for critically ill patients. Pain is harder to evaluate in non-communicative patients, who can´t report their own pain. Behavioral indicators have been proved as useful and reliable for detecting and measuring pain in these patients, and have been the basis for constructing scales for measuring pain, such as the Behavioural Pain Scale (BPS), the Critical Care Observation Tool (CPOT) and the Scale of Behaviors Indicating Pain (ESCID) .

The BPS and ESCID were tested in a study with a sample of 42 critically ill patients in Spain, showing good validity and reliability.

The objective of this Spanish multicentre study is to test the validity and reliability of the ESCID scale in a large sample of critically ill patients with medical and postsurgical pathology for the detection and measurement of pain.

DETAILED DESCRIPTION:
The specific Aims for the study are :

To determine the validity and reliability of the ESCID scale to assess pain in non-communicative critically ill patients on mechanical ventilation, in a large sample of critically ill medical and surgical patients.

To assess the relationship between the application of a common and painful procedure, usual in daily practice, and its associated changes in physiological indicators of pain: variation of heart rate, blood pressure, respiratory rate, sweating.

To assess the degree of pain when applying two painful procedures documented as common in the usual care of critically ill patients, and one non-painful procedure, using two pain scales: ESCID and BPS.

To assess the differences in the employment of the pain scales in patients with medical and surgical pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older
* Patient's primary language spanish where the evaluation is performed
* Patient meets IRB/Central EC requirements of the institution/ country where the evaluation is performed
* Patient is receiving the study's procedures as part of standard care, excepting the non painful procedure

Exclusion Criteria:

* Patient's condition is very unstable at the time of measurement of pain
* Patient is receiving neuromuscular blocking medications at the time of measurement of pain
* Patient´s probable or diagnosed delirium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients who are uncommunictive, receiving mechanical ventilation and undergoing any of the study procedures. Consent to participate will be requested to the family of the patient. Adults age 18 and over will be eligible for the study if they meet study inclusion criteria and don't meet any exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 20 minutes
  Pain intensity will be measured through the use of 2 scales based on behaviour items, the Behavioural Pain Scale (BPS) and the ''Scale of Behavioral Indicators of Pain'' (ESCID-Escala de Conductas Indicadoras de Dolor), by two independent observers with blind result among them, when the application of two procedures registered as painful (PD) and common in clinical practice, mobilization and tracheal suctioning, and one non-painful procedure (PND). The measurement will be performed once per each patient and procedure. The measurement of pain will be carried out in 3 stages: 5 minutes before the PD/PND, during PD/PND and 15 minutes after PD/PND.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Latorre, RN, Principal Investigator — Puerta de Hierro Majadahonda University Hospital. Medical ICU. Spain.
Locations (1):
- Puerta de Hierro Majadahonda University Hospital. Intensive Care Unit., Majadahonda, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Latorre-Marco I, Solis-Munoz M, Acevedo-Nuevo M, Hernandez-Sanchez ML, Lopez-Lopez C, Sanchez-Sanchez Mdel M, Wojtysiak-Wojcicka M, De las Pozas-Abril J. Validation of the Behavioural Indicators of Pain Scale ESCID for pain assessment in non-communicative and mechanically ventilated critically ill patients: a research protocol. J Adv Nurs. 2016 Jan;72(1):205-16. doi: 10.1111/jan.12808. Epub 2015 Sep 11. PMID 26358885
- [Result] Latorre-Marco I, Acevedo-Nuevo M, Solis-Munoz M, Hernandez-Sanchez L, Lopez-Lopez C, Sanchez-Sanchez MM, Wojtysiak-Wojcicka M, de Las Pozas-Abril J, Robleda-Font G, Frade-Mera MJ, De Blas-Garcia R, Gorgolas-Ortiz C, De la Figuera-Bayon J, Cavia-Garcia C. Psychometric validation of the behavioral indicators of pain scale for the assessment of pain in mechanically ventilated and unable to self-report critical care patients. Med Intensiva. 2016 Nov;40(8):463-473. doi: 10.1016/j.medin.2016.06.004. Epub 2016 Aug 31. English, Spanish. PMID 27590592